CLINICAL TRIAL: NCT06827600
Title: The Effect of Breastfeeding Training Given to Nulliparous Pregnant Women Before Cesarean Section on Breastfeeding Intention and Attitudes in the Postpartum Period: A Randomized Controlled Trial
Brief Title: Breastfeeding Intention and Breastfeeding Attitudes in the Postpartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gonca Buran, PhD, RN, Assit. Prof., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 915
Record Dates: First submitted 2025-01-27; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Caesarean Section; Nulliparous; Breastfeeding, Exclusive; Breastfeeding Attitude
Keywords: Caesarean section; Nulliparous; Breastfeeding, Exclusive; Breastfeeding attitude; Breastfeeding intention
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: Following recruitment, the pregnant women were divided into a study and a control group by randomization (1:1 randomization)
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The Care Provider and Outcome Assessor will be kept unaware of the experimental and control groups participating in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The experimental group in this study received structured breastfeeding education in addition to the standard care provided by healthcare professionals.
  Interventions: Behavioral: Structured breastfeeding education and follow-up
- Control group (No Intervention): The control group was in the usual care.

INTERVENTIONS:
Behavioral: Structured breastfeeding education and follow-up — Breastfeeding education was provided face-to-face to mothers assigned to the experimental group. The authors developed a breastfeeding education program and prepared a booklet. This booklets were distributed to experimental group.Follow-up were carried out on the 3rd day and at the 1st, 3rd, and 6th months postpartum. each follow-up session, the educational program's core components were reinforced through a standardized summary, ensuring continuity and clarity in the information provided.
  Training Content
  * Significance of Breastfeeding
  * Advantages of Breastfeeding
  * Overview of Colostrum
  * Duration for Breastfeeding
  * Breastfeeding Positions
  * Strategies for Enhancing Breast Milk Production
  * Increasing Breast Milk Supply
  * Techniques for Placing the Baby on the Breast
  * Implications of Improper Baby Positioning
  * Indicators of Sufficient Breast Milk for the Infant
  * Expressing Breast Milk
  * Recommendations for Storing Expressed Milk
  Arms: Experimental group

SUMMARY:
Purpose:

It will be carried out to determine the effect of breastfeeding education given to nulliparous pregnant women before cesarean section on breastfeeding intention and breastfeeding attitudes in the postpartum period.

Material method:

The research, planned as a randomized controlled experimental study, will be carried out with a total of 70 mothers who are hospitalized in the Maternity Clinic of Bursa Uludağ University Research and Practice Hospital and who meet the study assignment criteria and who are determined by simple randomization method. Breastfeeding education and support will be provided to 35 women in the experimental group, and 35 women in the control group will be left to the hospital's usual care. Data will be collected between April 2024 and January 2025 using the "Introductory Form," "Newborn Feeding Intention Scale," and "Breastfeeding Attitude Evaluation Scale." The educational intervention will be carried out one-on-one in the woman's own room during the prenatal period for the women allocated to the experimental group. In addition to the explanation, question and answer, and visual material use, the demonstration technique with a newborn model will be used in the education. A booklet containing written illustrated breastfeeding education prepared in line with the literature will be given to mothers with cesarean delivery. The data will be filled in the "Introductory Information Form," "Newborn Feeding Intention Scale," and "Breastfeeding Attitude Assessment Scale." The data of the study will be analyzed in the Statistical Package for the Social Sciences (SPSS) for Windows 20.0 package program. Descriptive statistics (arithmetic mean, minimum-maximum, standard deviation, number, and percentage), Student t-test, one-way analysis of variance (ANOVA), Mann-Whitney U test, and Kruskal-Wallis test will be used in the analysis of the data.

Expected Result:

Determining the effect of breastfeeding education given to nulliparous pregnant women before cesarean section on breastfeeding intention and breastfeeding attitudes in the postpartum period will guide health professionals. It will be a resource for studies that can be conducted on different sample groups and in different regions on the subject and will contribute to national and international literature and scientific knowledge with the publication to be made.

DETAILED DESCRIPTION:
Cesarean section rates are increasing every year worldwide and in Turkey. Due to the effects of anesthesia and pain in the cesarean area, breastfeeding and continuing breastfeeding are difficult. Breastfeeding is very important for maintaining the healthy growth of newborns, preventing future health problems such as obesity and cardiovascular diseases, and for maternal health. For these reasons, the World Health Organization (WHO) recommends that babies be fed only breast milk for the first six months and that breastfeeding should continue for two years.

Data from the Organization for Economic Co-operation and Development (OECD) indicate that numerous countries have cesarean section rates that surpass the recommended thresholds. Notably, Turkey has the highest cesarean section rate at 53.1%. Research has demonstrated that cesarean deliveries can pose challenges in initiating and sustaining breastfeeding.

Achieving WHO's 2030 goals on breast milk and breastfeeding, increasing breast milk intake, and increasing breastfeeding rates at the national level will directly contribute to maternal and child health and indirectly reduce family and health expenditures. However, when previous studies in the literature are examined, it is known that cesarean births, the effects of anesthesia, and pain in the cesarean area make breastfeeding and continuing breastfeeding a difficult factor.

This research project, which is planned as a randomized controlled experimental study, will be carried out to determine the effect of breastfeeding education and support given to nulliparous pregnant women before cesarean on breastfeeding intentions and breastfeeding attitudes in the postpartum period.

Research Questions:

1. Is there a difference between the breastfeeding intentions of women in the experimental and control groups before the education intervention?
2. Is there a difference between the breastfeeding intentions of women in the experimental and control groups after the education intervention?
3. Is there a difference between the time when women who received breastfeeding education and support and women who did not receive it started breastfeeding?
4. Is there a difference in the attitudes of women who received breastfeeding education and support and those who did not receive cesarean section regarding breastfeeding in the postpartum period?
5. 5. Is there a difference in the delivery times between women who receive breastfeeding education and support and those who do not?

The project aims to ensure that mothers who gave birth by cesarean section and were given breastfeeding education and support will feed their babies exclusively with breast milk for at least 6 months to continue their breastfeeding intention and breastfeeding attitude and to increase the breastfeeding rates of mothers who gave birth by cesarean section.

Target measurements

* Before and after education (while pregnant before cesarean section)
* During discharge (postpartum period),
* In the first, third, and sixth months after discharge, the process will be conducted by phone call.

It aims to analyze and report the results of the newborn breastfeeding duration intention and breastfeeding attitude scale scores of the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older,
* Speaking and understanding Turkish,
* Having a planned Caesarean section,
* Being nulliparous

Exclusion Criteria:

* Having a history of psychological or mental health problems
* Having any condition in the mother or infant that was a barrier to breastfeeding (using medication that passes into breast milk, breast structure not being suitable for milk production, mastectomy operation, etc.)
* The baby's admission into the neonatal unit
* The baby's separation from the mother for any reason
* Having a disease (anomaly, cleft palate and lip, etc.) that prevents the baby from breastfeeding,
* Having given childbirth outside of the 37-42nd week,
* Having a baby with a birth weight below 2500 grams

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Infant feeding Intentions before Intervention | before Intervention (37th and 42nd weeks of pregnancy)
  Before the breastfeeding education intervention, the "Infant Feeding Intentions Scale" was applied to the pregnant women in the experimental and control groups. The intentions of the pregnant women in both groups to breastfeed their babies were evaluated.According to the score of the Infant Feeding Intentions Scale, breastfeeding intention is classified as follows: (0-3.5) very low, (4.0-7.5) low, (8.0-11.5) moderate, (12.0-15.5) strong and (16.0) very strong.
Breastfeeding intentions after Intervention | after Intervention (37th and 42nd weeks of pregnancy)
  After the breastfeeding education intervention in the experimental group, the "Infant Feeding Intentions Scale" was applied to the pregnant women in the experimental and control groups. The intentions of both groups to breastfeed their babies were determined.groups. The intentions of the pregnant women in both groups to breastfeed their babies were evaluated.According to the score of the Infant Feeding Intentions Scale, breastfeeding intention is classified as follows: (0-3.5) very low, (4.0-7.5) low, (8.0-11.5) moderate, (12.0-15.5) strong and (16.0) very strong.
Breastfeeding intentions before discharge | Postpartum 3rd day
  Before discharge, mothers in both the experimental and control groups were administered the "Infant Feeding Intentions Scale". The intentions of the mothers in both groups to breastfeed their babies were evaluated. According to the score of the Infant Feeding Intentions Scale, breastfeeding intention is classified as follows: (0-3.5) very low, (4.0-7.5) low, (8.0-11.5) moderate, (12.0-15.5) strong and (16.0) very strong. As the score of the breastfeeding attitude scale increases, it is evaluated that the breastfeeding attitude is positive. The scale has no subgroups.
Breastfeeding attitude before discharge | Postpartum 3rd day
  Before discharge, mothers in both the experimental and control groups were administered the "Breastfeeding Attitude Scale." This instrument yields scores ranging from 0 to 184, with one item being reverse-scored. An increase in the score reflects a more positive attitude toward breastfeeding.
Breastfeeding intentions: postpartum 1st month | Postpartum 1st month
  The mothers in the experimental and control groups were assessed using the "Infant Feeding Intentions Scale" on the first month postpartum. According to the score of the Infant Feeding Intentions Scale, breastfeeding intention is classified as follows: (0-3.5) very low, (4.0-7.5) low, (8.0-11.5) moderate, (12.0-15.5) strong and (16.0) very strong. As the breastfeeding attitude scale scores increase, it is evaluated that the breastfeeding attitude is positive. The scale has no subgroups.
Breastfeeding attitude: postpartum 1st month | Postpartum 1st month
  The mothers in the experimental and control groups were assessed using the "Breastfeeding Attitude Assessment Scale" during the first month postpartum. This instrument yields scores ranging from 0 to 184, with one reverse-scored item. An increase in the score reflects a more positive attitude toward breastfeeding.
Breastfeeding Intentions: postpartum 3rd month | Postpartum 3rd month
  The mothers in the experimental and control groups were assessed using the "Infant Feeding Intentions Scale" on the 3rd month postpartum. According to the score of the Infant Feeding Intentions Scale, breastfeeding intention is classified as follows: (0-3.5) very low, (4.0-7.5) low, (8.0-11.5) moderate, (12.0-15.5) strong and (16.0) very strong. As the breastfeeding attitude scale scores increase, it is evaluated that the breastfeeding attitude is positive. The scale has no subgroups.
Breastfeeding attitude: postpartum 3rd month | Postpartum 3rd month
  The mothers in the experimental and control groups were assessed using the "Breastfeeding Attitude Assessment Scale" during the 3rd month postpartum. This instrument yields scores ranging from 0 to 184, with one reverse-scored item. An increase in the score reflects a more positive attitude toward breastfeeding.
Breastfeeding Intentions: postpartum 6th month | Postpartum 6th month
  The mothers in the experimental and control groups were assessed using the "Infant Feeding Intentions Scale" on the 6th month postpartum. According to the score of the Infant Feeding Intentions Scale, breastfeeding intention is classified as follows: (0-3.5) very low, (4.0-7.5) low, (8.0-11.5) moderate, (12.0-15.5) strong and (16.0) very strong. As the breastfeeding attitude scale scores increase, it is evaluated that the breastfeeding attitude is positive. The scale has no subgroups.
Breastfeeding attitude: postpartum 6th month | Postpartum 6th month
  In the 6th month postpartum, mothers in both the experimental and control groups underwent evaluation using the "Breastfeeding Attitude Assessment Scale." This scale generates scores ranging from 0 to 184, with one item scored in reverse. An increase in the total score signifies a more positive attitude toward breastfeeding.

SECONDARY OUTCOMES:
The starting breastfeeding in the first hour | Postpartum 3rd day
  Assessed using the Breastfeeding Follow-up Form in 3rd day postpartum. Mothers reported whether they started breastfeeding within the first hour after birth
Bottle feeding | Postpartum 3rd day
  Assessed using the Breastfeeding Follow-up Form in 3rd day postpartum. Mothers reported whether they started breastfeeding within the first hour after birth.
  Mothers reported whether they feed her baby with exclusively mother's milk.
Exclusively feeding with mother's milk | postpartum 1sth month
  Breastfeeding was assessed using the Breastfeeding Follow-up Form. Mothers provided information regarding whether they practiced exclusive breastfeeding during the first month following the birth of their child.
  Mothers reported whether they feed her baby with exclusively mother's milk.
Exclusively feeding with mother's milk | Postpartum 3rd month
  Breastfeeding was assessed using the Breastfeeding Follow-up Form. Mothers provided information regarding whether they practiced exclusive breastfeeding during the 3rd month following the birth of their child.
Exclusively feeding with mother's milk | Postpartum 6th month
  Breastfeeding was assessed using the Breastfeeding Follow-up Form. Mothers provided information regarding whether they practiced exclusive breastfeeding during the 6th month following the birth of their child.

CONTACTS AND LOCATIONS:
Overall Officials: Gonca Buran, Principal Investigator — Uludag University
Locations (1):
- Uludag University, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Güneri, S. E., Muslu, G. K., & Güner, Ö. (2019). The Turkish Version of the Infant Feeding Intention Instrument (IFI-T). 41(3): 269-74
- [Background] Buran G, Ozyazicioglu N, Aydin AI, Atak M. Evaluation of breastfeeding success and self-efficacy in mothers giving birth via vaginal delivery or cesarean section: a cross-sectional study. Women Health. 2022 Oct-Dec;62(9-10):788-798. doi: 10.1080/03630242.2022.2146832. Epub 2022 Nov 20. PMID 36404416
- [Result] Hobbs AJ, Mannion CA, McDonald SW, Brockway M, Tough SC. The impact of caesarean section on breastfeeding initiation, duration and difficulties in the first four months postpartum. BMC Pregnancy Childbirth. 2016 Apr 26;16:90. doi: 10.1186/s12884-016-0876-1. PMID 27118118
- [Result] Li L, Wan W, Zhu C. Breastfeeding after a cesarean section: A literature review. Midwifery. 2021 Dec;103:103117. doi: 10.1016/j.midw.2021.103117. Epub 2021 Aug 14. PMID 34425257